CLINICAL TRIAL: NCT06433206
Title: Quality of Life, Symptom Severity, and Care Needs in Lung Cancer Patients Receiving Immunotherapy
Brief Title: Care Needs in Lung Cancer Patients Receiving Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201911078RIND
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer, Immunotherapy, Quality of Life, Symptom Severity, Care Needs
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Lung cancer ranks as the leading cause of cancer-related deaths globally and is among the most common malignancies. In recent years, the advancements in immune checkpoint inhibitors have marked a significant breakthrough in the immunotherapy of lung cancer. However, immunotherapy is a relatively new treatment modality, and ongoing clinical trials continue to explore its efficacy. Due to a lack of knowledge about immunotherapy-related care, patients often experience uncertainty and anxiety regarding its effectiveness, resulting in associated care needs.

A total of 160 lung cancer patients were included in the study. The research findings revealed statistically significant correlations (p < 0.05) between the severity of disease, symptomatology, overall health status, functional capacity, cognitive function, disease progression, mood, and general supportive care needs, as well as specific needs of lung cancer patients.

Regarding factors influencing care needs, it was found that general supportive care needs were significantly influenced by marital status, average personal monthly income, and disease progression. Additionally, age, surgical history, functional capacity, and cognitive function significantly influenced specific care needs. Based on these statistical findings, it is crucial for nursing staff to closely monitor changes in patients' symptoms and mood and provide timely care and support. Furthermore, future interventions should focus on addressing the heightened needs of lung cancer patients, thereby reducing their dissatisfaction along the cancer treatment journey.

DETAILED DESCRIPTION:
Background and Purpose: Lung cancer is a major health concern affecting the Taiwanese population. Immunotherapy represents a novel treatment approach which activates the immune system to combat tumor cells through a series of interactions. However, the side effects associated with immunotherapy can be significant, potentially causing uncertainty and anxiety in patients. Medical decision-making also involves numerous considerations, impacting their psychosocial well-being and subsequent health behaviors. Research in this area remains limited. Therefore, this study aims to (1) explore the quality of life, severity of symptoms, and care needs of lung cancer patients following immunotherapy; (2) investigate the correlations between quality of life, severity of symptoms, and care needs; and (3) identify predictive factors for the care needs of immunotherapy patients.

Research Method: This study adopts a cross-sectional research design, conducted at a medical center and a specialized cancer hospital in Taipei City. Recruitment takes place in hospital wards, treatment rooms, and outpatient clinics, utilizing consecutive sampling. Lung cancer patients who have undergone or are currently undergoing immunotherapy are selected. Structured questionnaires are employed, covering demographics, disease treatment characteristics, severity of symptoms, quality of life, functional disability, supportive care needs, fear of disease progression, and qualitative interviews. Quantitative data are analyzed using descriptive and inferential statistics in SPSS version 22.0. The study aims to enroll 180 participants.

Expected Results: The anticipated findings of this study are expected to provide valuable insights for clinical healthcare professionals. They can aid in understanding patients' needs, contribute to the development of post-immunotherapy care guidelines for lung cancer patients, and serve as essential references for healthcare reimbursement policies. These outcomes may help alleviate patient burden and enhance quality of life. It is expected that demographic characteristics, disease treatment characteristics, quality of life, severity of symptoms, and the extent of care needs will be positively correlated and serve as important predictors of care needs.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with malignant lung tumors based on imaging or post-surgical histopathological examination results by specialized physicians.
2. Individuals who have received immunotherapy in the past or are currently undergoing immunotherapy.
3. Research participants who are conscious, aged 20 years or older, able to communicate in Mandarin or Taiwanese, capable of completing the questionnaire, willing to participate in the study, and have signed the research consent form.

Exclusion Criteria:

1. Individuals with significant cognitive impairments who are unable to complete the questionnaire.
2. Individuals who are unable to communicate in Mandarin or Taiwanese.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using consecutive sampling, lung cancer patients who have received or are currently undergoing immunotherapy will be selected from a medical center and a specialized cancer hospital in northern Taiwan.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Care Needs in Lung Cancer Patients Receiving Immunotherapy | 1year

SECONDARY OUTCOMES:
Quality of Life in Lung Cancer Patients Receiving Immunotherapy | 1year
Symptom Severity in Lung Cancer Patients Receiving Immunotherapy | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ping Hsiao, master, Principal Investigator — NTUCC
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan